CLINICAL TRIAL: NCT06084078
Title: Patient Identification, Prescreening and LDCT Screening for Lung Cancer With Telehealth
Brief Title: Rural Illinois Lung Cancer Screening Initiative
Acronym: LDCT
Status: Not yet recruiting | Type: Observational
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Other Study IDs: LDCT Screening
Record Dates: First submitted 2023-09-27; First posted 2023-10-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
Keywords: cancer screening; LDCT; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telehealth cohort: Individuals who opt to do the screening using telehealth. Telehealth using video assisted techniques or using telephone.
- In-person cohort: Individuals who are willing to travel to the hospital for in-person screening and follow-up

SUMMARY:
The role of this observational study is to access the feasibility of providing lung cancer screening using a designated nurse navigator through lung cancer screening clinic. Eligible participants will be identified using medical records, eligibility will be confirmed through phone call, screening visits will be scheduled as in-person visit or telehealth visit. Computed tomography screening will be performed at an approved center closer to the individuals place of living and results will be discussed during follow-up in-person visit or telehealth visit.

DETAILED DESCRIPTION:
The long-term goal is to establish healthcare practices to increase adherence to lung cancer screening among high-risk individuals. The overall objective in this application is to establish a lung cancer screening initiative to proactively identify and screen eligible patients for LDCT using a designated nurse practitioner (NP) along with telehealth. The central hypothesis is that use of a designated NP along with telehealth will increase lung cancer screening via LDCT among high-risk, racial/ethnic minority, and rural/sub-urban patients. The rationale for this proposal is use of a NP and telehealth will help overcome the barriers physicians face in identifying eligible patients for LDCT including collecting additional information to determine eligibility, discussing the pros and cons of LDCT, providing smoking cessation/abstinence counseling, making shared decisions, and documenting this information in the patients' charts.

In this prospective cohort study the nurse practitioner (NP) will proactively identify eligible individuals for LDCT using EMRs that are shared across the Department of Family and Community Medicine at SIU. These patients will be contacted and those agreeing to undergo screening will be given a referral to a nearby LDCT center. The NP will follow-up with the patients with the results of the LDCT and will refer them for further management to their primary care physician. If the results are negative for nodules then they will be followed up on a yearly basis until the participants are older than 80 years or have other life-threatening health issues.

ELIGIBILITY:
Inclusion Criteria:

* All individuals 50-80 years of age
* 20 pack-year smoking history
* Currently smoke or have quit within the past 15 years:

Exclusion Criteria:

* Individuals 49 years and below or 81 years and above
* Has not smoked in 15 or more years
* Individuals who develop a health problem that makes them unwilling or unable to have surgery if lung cancer is detected.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The risk of lung cancer increases with age and smoking status and hence this age range is recommended for receiving lung cancer screening. As per USPSTF criteria our screening initiative will include individuals 50-80 years, subjects of all sex/gender and all race/ethnic groups. Screening eligible individuals included in our pilot study consisted of 54.4 % women, 75% of non-Hispanic whites, 24% non-Hispanic blacks and 1.2% belonged to 'other' race category. Non-Hispanic black individuals with smoking history have a higher risk of developing lung cancer than a non-Hispanic white. Very few Hispanic persons and women tend to accumulate fewer pack-years over a long period of time.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Screening rate | Through study completion, an average of 1 year
  Percentage of individuals screened (completed CT imaging) with and without telehealth
Early stage diagnosis | Through study completion, an average of 1 year
  Percentage of individuals diagnosed with lung cancer at an early stage of the disease

SECONDARY OUTCOMES:
Time to treatment initiation | Through study completion, an average of 1 year
  Number of days from diagnosis to treatment initiation will be calculated for each patient diagnosed with lung cancer
Adherence to Screening | Through study completion, an average of 1 year
  Percentage of of individuals undergoing yearly screening with and without telehealth
Cost | Through study completion, an average of 1 year
  Overall cost from pre-screening to screening and follow-up with and without telehealth

CONTACTS AND LOCATIONS:
Overall Officials: Sowmy Thuppal, MD PhD, Principal Investigator — Southrn Illinois University School of Medicine

IPD SHARING:
Plan to Share IPD: No
The goal of this project is to look a at telehealth vs in-person screening. Overall aggregates will be shared with the scientific community to assess if telehealth is a better option for screening.

REFERENCES:
- [Result] Thuppal S, Hendren JR, Colle J, Sapra A, Bhandari P, Rahman R, Krus-Johnston A, Hoffman MR, Foray N, Hazelrigg S, Crabtree T. Proactive Recruitment Strategy for Patient Identification for Lung Cancer Screening. Ann Fam Med. 2023 Mar-Apr;21(2):119-124. doi: 10.1370/afm.2905. PMID 36973046
- [Result] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641